CLINICAL TRIAL: NCT01101854
Title: Gene Expression Profiles in Healing and Non-Healing Wounds
Acronym: GeneScreen
Status: Terminated | Type: Observational
Why Stopped: PI left Indiana University and has elected not to continue this project at new institution.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Gayle Gordillo, Professor, Indiana University
Other Study IDs: 1906520102; NCT00618189 (obsolete NCT alias)
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-02

CONDITIONS: Wounds and Injuries
Keywords: gene expression in wounds; healing wounds; non-healing wounds; punch biopsy; debridement
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to develop a database containing information about genes/proteins/fats as well as wound infections in both healing and non-healing wounds. Many wounds that do not heal are infected. This study will help us determine if there is a relationship between the types of infections and how well a wound heals. Identification of genes/proteins/lipids (fats) that help predict wound healing under specific wound healing conditions will enable health care practitioners to select more appropriate treatments, monitor the responses to those treatments, and figure out what standard treatments should be.

DETAILED DESCRIPTION:
During the first study visit, information about participants, such as age, race and gender, medical history, including nutritional status, medications and dietary supplements, and genetic diseases in the participant's family will be collected. Smoking and tobacco status, alcohol consumption, and/or recreational drugs usage will be documented. Additionally, wound information, including wound measurements, infection history, cause, location, how long you have had the wound, etc, a digital photograph of the wound and ultrasound imaging (if available) will be obtained. Lab results, such as nutrition and blood sugar (if the subject has Diabetes Mellitus) levels will be obtained. If a blood sugar level is not available from the past 3 months, a finger stick will be performed to obtain the participant's hemoglobin A1c level. Lastly, debrided tissue and/or biopsies, wound fluid, and 20 cc of blood will be collected.

During second study visit, a digital image of the wound area will be taken and the wound will be evaluated for clinical signs of infection using a WIfI scale, as appropriate. Any new wound treatments, labs, and adverse events along with changes in medications and medical history since baseline will be documented. Additionally, debrided tissue and/or biopsies, wound fluid, and 20 cc of blood will be collected.

The final stage is the observation phase, which will last up to 12 weeks. The wound closure and/or area data will be recorded from the participant's medical record up to 12 weeks.

Potential Risks:

Biopsy and Debridement:

There may be some discomfort with the tissue biopsy procedure depending on the amount of sensation the subject has at the site of the wound. The wound site will be numbed by applying local anesthesia as appropriate to area being biopsied. The amount of pain that occurs with wound biopsy will vary from person to person, but all reasonable efforts will be made to minimize pain. The biopsy procedure is done within the boundaries of the existing wound to avoid giving the patient a separate new wound. Bleeding is a possible complication, but the risk is low for the small biopsies and is reduced by using local anesthetics with epinephrine, and silver nitrate sticks are available in each room to cauterize biopsy sites as needed. Infection is also a potential risk; however, wound tissue biopsies are routinely performed as the standard of care in the CWC to diagnose wound infection. The biopsy site will be appropriately monitored for infection by the provider managing the wound during routine wound clinic visits. No additional study specific risk is identified for debrided tissue as the procedure is performed as part of SoC.

Blood Draw:

Temporary discomfort from the needle stick, bruising, bleeding, and rarely, infection. To reduce the risk of infection, the research personnel will clean subject's arm with an antiseptic solution before any blood is drawn.

Hemoglobin A1c point-of-care testing:

The point-of-care testing for hemoglobin A1c test is low risk. Potential risks include minor and temporary pain or discomfort and bleeding. Prior to the finger prick, research staff will clean the finger to be pricked with an alcohol swab. Subjects will be provided with a cotton ball and/or band-aid to stop the bleeding, if there is any.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and above
* Ulcer duration of > 4 weeks

Exclusion Criteria:

* Pregnant females
* Receiving chemotherapy or radiation therapy for cancer
* Known or suspected malignancy of current study ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a chronic wound(s) (defined as a wound that has been present for at least 4 weeks).
Sampling Method: Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-10-23 (Actual); Study Completion 2021-10-23 (Actual)

PRIMARY OUTCOMES:
Gene Expression Profiles | 12 weeks
  A database of gene/protein/lipid expression and wound infection in healing and non-healing wounds.

SECONDARY OUTCOMES:
Wound microbiome in healing and non-healing wounds | 12 weeks
  Identify the difference in microbiome between healing and non-healing wounds.
Wound area at baseline vs 12 weeks | 12 weeks
  Compare the wound area during baseline visit and 12 weeks later.
Ultrasound images (per availability) | 12 weeks
  Capture ultrasound images to understand anatomical nature of healed and non-healing wounds.
Histopathological analysis in healing vs non-healing wounds | 12 weeks
  Compare the differences in tissue from healing and non-healing wounds.

CONTACTS AND LOCATIONS:
Overall Officials: Gayle Gordillo, MD, Principal Investigator — Indiana University
Locations (1):
- IU Health Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meehan M, O'Hara L, Morrison YM. Report on the prevalence of skin ulcers in a home health agency population. Adv Wound Care. 1999 Nov-Dec;12(9):459-67. PMID 10687558
- [Background] Pieper B, Templin TN, Dobal M, Jacox A. Wound prevalence, types, and treatments in home care. Adv Wound Care. 1999 Apr;12(3):117-26. PMID 10655791
- [Background] Gottrup F, Holstein P, Jorgensen B, Lohmann M, Karlsmar T. A new concept of a multidisciplinary wound healing center and a national expert function of wound healing. Arch Surg. 2001 Jul;136(7):765-72. doi: 10.1001/archsurg.136.7.765. PMID 11448387
- [Background] Coerper S, Wicke C, Pfeffer F, Koveker G, Becker HD. Documentation of 7051 chronic wounds using a new computerized system within a network of wound care centers. Arch Surg. 2004 Mar;139(3):251-8. doi: 10.1001/archsurg.139.3.251. PMID 15006880
- [Background] Kalani M, Brismar K, Fagrell B, Ostergren J, Jorneskog G. Transcutaneous oxygen tension and toe blood pressure as predictors for outcome of diabetic foot ulcers. Diabetes Care. 1999 Jan;22(1):147-51. doi: 10.2337/diacare.22.1.147. PMID 10333917
- [Background] Grolman RE, Wilkerson DK, Taylor J, Allinson P, Zatina MA. Transcutaneous oxygen measurements predict a beneficial response to hyperbaric oxygen therapy in patients with nonhealing wounds and critical limb ischemia. Am Surg. 2001 Nov;67(11):1072-9; discussion 1080. PMID 11730224
- [Background] Misuri A, Lucertini G, Nanni A, Viacava A, Belardi P. Predictive value of transcutaneous oximetry for selection of the amputation level. J Cardiovasc Surg (Torino). 2000 Feb;41(1):83-7. PMID 10836229
- [Background] Niinikoski J. Hyperbaric oxygen therapy of diabetic foot ulcers, transcutaneous oxymetry in clinical decision making. Wound Repair Regen. 2003 Nov-Dec;11(6):458-61. doi: 10.1046/j.1524-475x.2003.11610.x. PMID 14617286
- [Background] Padberg FT, Back TL, Thompson PN, Hobson RW 2nd. Transcutaneous oxygen (TcPO2) estimates probability of healing in the ischemic extremity. J Surg Res. 1996 Feb 1;60(2):365-9. doi: 10.1006/jsre.1996.0059. PMID 8598670
- [Background] Gordillo GM, Schlanger R, Wallace WA, Bergdall V, Bartlett R, Sen CK. Protocols for topical and systemic oxygen treatments in wound healing. Methods Enzymol. 2004;381:575-85. doi: 10.1016/S0076-6879(04)81037-1. No abstract available. PMID 15063699
- [Background] Patterson JA, Bennett RG. Prevention and treatment of pressure sores. J Am Geriatr Soc. 1995 Aug;43(8):919-27. doi: 10.1111/j.1532-5415.1995.tb05538.x. No abstract available. PMID 7636103
- [Background] Roy S, Rink C, Khanna S, Phillips C, Bagchi D, Bagchi M, Sen CK. Body weight and abdominal fat gene expression profile in response to a novel hydroxycitric acid-based dietary supplement. Gene Expr. 2004;11(5-6):251-62. doi: 10.3727/000000003783992289. PMID 15200237
- [Background] Roy S, Khanna S, Wallace WA, Lappalainen J, Rink C, Cardounel AJ, Zweier JL, Sen CK. Characterization of perceived hyperoxia in isolated primary cardiac fibroblasts and in the reoxygenated heart. J Biol Chem. 2003 Nov 21;278(47):47129-35. doi: 10.1074/jbc.M308703200. Epub 2003 Sep 2. PMID 12952964
- [Background] Roy S, Lado BH, Khanna S, Sen CK. Vitamin E sensitive genes in the developing rat fetal brain: a high-density oligonucleotide microarray analysis. FEBS Lett. 2002 Oct 23;530(1-3):17-23. doi: 10.1016/s0014-5793(02)03309-4. PMID 12387859
- [Background] Roy S, Khanna S, Bentley K, Beffrey P, Sen CK. Functional genomics: high-density oligonucleotide arrays. Methods Enzymol. 2002;353:487-97. doi: 10.1016/s0076-6879(02)53071-8. No abstract available. PMID 12078521
- [Background] Liu-Stratton Y, Roy S, Sen CK. DNA microarray technology in nutraceutical and food safety. Toxicol Lett. 2004 Apr 15;150(1):29-42. doi: 10.1016/j.toxlet.2003.08.009. PMID 15068823
- [Background] Eisen MB, Spellman PT, Brown PO, Botstein D. Cluster analysis and display of genome-wide expression patterns. Proc Natl Acad Sci U S A. 1998 Dec 8;95(25):14863-8. doi: 10.1073/pnas.95.25.14863. PMID 9843981
- [Background] Pawitan Y, Michiels S, Koscielny S, Gusnanto A, Ploner A. False discovery rate, sensitivity and sample size for microarray studies. Bioinformatics. 2005 Jul 1;21(13):3017-24. doi: 10.1093/bioinformatics/bti448. Epub 2005 Apr 19. PMID 15840707
- [Background] Efron B, Tibshirani R, Storey JD, Tusher V. Empirical Bayes Analysis of a Microarray Experiment. Journal of the American Statistical Association. 2001; 96(456):1151-1160.